CLINICAL TRIAL: NCT04618926
Title: A Prospective Randomized Study Comparing Fiberoptic Bronchoscope Endotracheal Intubation Between the Intubating Laryngeal Tube Suction and the LMA Protector
Brief Title: A Comparison of Fiberoptic Endotracheal Intubation Between the Intubating Laryngeal Tube Suction and the LMA Protector
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, Associate Clinical Professor of Anesthesiology, Bnai Zion Medical Center
Other Study IDs: PROTECTOR
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Difficult Airway
Keywords: iLTS-D, LMA Protector, Fiberoptic intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- intubating Laryngeal Tube Suction Disposable: intubating Laryngeal Tube Suction Disposable Airway control
  Interventions: Device: Device intubating Laryngeal Tube Suction Disposable
- intubating laryngeal Tube suction Disposable: intubating laryngeal Tube Suction Disposable
  Interventions: Device: Device intubating Laryngeal Tube Suction Disposable

INTERVENTIONS:
Device: Device intubating Laryngeal Tube Suction Disposable — Resuscitation in covid 19 patients
  Other Names: Device LMA Protector

SUMMARY:
Securing the airway is a pivotal skill for anesthesiologists and emergency care providers. Endotracheal intubation (ETI) is considered the gold standard for securing the airway.

When ETI via laryngoscopy has failed, the use of a supraglottic airway device (SGAD) has been recommended. The intubating Laryngeal Tube Suction-Disposable and the LMA Protector are a new step in the evolution of supraglottic airways. Both SGADs are enable to ventilation and oxygenation, but the ventilation channel allow the insertion of an endotracheal tube and the use of fiberoptic bronchoscope. The aim of this study is to compare the time of fiberoptic intubation through the intubating Laryngeal Tube Suction Disposable and the LMA Protector in adult patients.

DETAILED DESCRIPTION:
Detailed Description: Securing the airway is a pivotal skill for anesthesiologist and emergency providers. Endotracheal intubation (ETI) is considered the gold standard for securing the airway. Induction time during anesthesia may sometimes present unexpected difficulties during ETI.

When ETI via laryngoscopy has failed, the use of a supraglottic airway device (SGAD) has been recommended. Previous studies suggested that compare intubation with laryngoscope, SGADs enables rapid and effective airway control. Improved second generation SGADs enable ventilation and oxygenation, but also include a second channel that separates the trachea from the esophagus preventing aspiration. According with the results of the Fourth National Audit Project of the Royal College of Anesthetist will bets and the Difficult Airway Society, the second generation SGADs should be uses instead the first generation.

Some of the second generations of SGADs have a ventilation channel that allow the insertion of an endotracheal tube.

Two of these devices recently introduced in the market are the intubating Laryngeal Tube Suction Disposable (iLTS-D) and the Laryngeal Mask Airway Protector [5, 6] The intubating Laryngeal Tube Suction- Disposable (iLTS-D) (VBM, Germany) is a new updated version of the Laryngeal Tube-Suction Disposable (LTS-D). [5] It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube (ETT) No 7.5 mm. for fiberoptic guidance. Similarly to the LTS-D, the iLTS-D also has a separate channel for gastric tubes placement up to a size of 18 Fr. The device is latex free, made of PVC, and like the original laryngeal tube (LT), can be inserted blindly.

The iLTS-D comes in one size. According to the depth of insertion, the device will be equivalent to size 4 for patients 175 to 190 cm tall, or size 5 for patients taller than 190 cm.

The LMA Protector™ Airway (Teleflex Ireland) will be a new step in the evolution of supraglottic airways. This is a single use device made mainly of silicone. The LMA Protector is designed to provide an opportunity to insert a tracheal tube of proper size through the device without the need of any special technique. [6] It is a PVC, double- lumen tube. One lumen will be used for ventilation and the others for gastric tube placement.

The ventilation channel has the ability to pass an ETT 7.5 mm with a fiberscope. The LMA Protector will be provide in sizes from 3, 4 and 5. The size 3 will be for patient of weight 30 to 50 Kg, the size 4 to patients of weight from 50 to 70 Kg and the size 5 to patients of weight 70 to 100 Kg.

Unlike the most of the second generation SGAD the LMA Protector possesses a shortand wide-bore preformed airway tube. Thwill be allows passage of wide internal diameter ETTs. It will be currently one of the few second-generation .SADs together with the iLTS-D that can also act as a conduit for endotracheal intubation.

The two SGDs will be inserted blindly with its distal tip positioned in the upper esophagus.

The aim of this be study will be to compare the time of fiberoptic intubation through the intubating Laryngeal Tube Suction Disposable and the LMA Protector in adult patients. The procedures will be performed by anesthesiologist with no previous experience with these two devices.

We hypothesized that the time needed for first-attempt successful fiberoptic-guided intubation with the two novel SADs would not differ by more than 10 s.

MATERIALS AND METHODS The study will obtain the approval of the Bnai Zion Medical Center Clinical Research Ethics Committee and will be obtain the registration from the ClinicalTrials.gov We will recruit patients if they have ≥18 years of age and of American Society of Anesthesiologic (ASA) physical status 1-2. Exclusion criteria included patients who have predicted to a difficult airway, who has any contraindication to the use of an SAD, weight > 90 Kg, aspiration risk and pregnancy woman.

After written informed consent , patients will be assigned, using a computer-generated randomized list, to having their airway intubated fibreopticaly through either an LMA Protector or iLTS-D. Patients will be blinded as to their allocation group.

The intubation will be performed by two experienced anesthesiologist, defined as having more than 10 years of clinical experience since the commencement of specialty and expert with Supraglottic Devices and fiberscope intubation.

All anesthesiologist involved in this study will participate in a standardized educational program and practice on an airway manikin and patients. Anesthesiologist will completed >10 uses on each device prior to the study either in simulators and patients.

The size of the LMA Protector was chosen by the intubating anesthesiologist based on the patient's weight and airway assessment. Size 3 to patient weighs of 30 to 50 Kg and size 4 to patient weight of 50 to 70 Kg. and 5 to patient weight of 70 to 100 Kg. The iLTS-D has only one size with marks in the proximal end of the device with the number 4 or 5 in order to guide the insertion more deep or more superficial according with the height of the patients. Number 4, color red, to adult height of 155-180 cm and number 5, color purple, to adult height of > 180 cm.

For each participant the following data will be recorded preoperatively: age, sex, height, weight, ASA physical status, predictors for difficult airway (Mallampati score, thyromental distance), and type of surgery.

After 3 minutes of pre-oxygenation with 100% oxygen to reach an end-tidal O2 ≥70 %, patients will be given induction agents.

Anesthesia will be induced with up to 2-3 mg/kg propofol, 3mcg/kg fentanyl and maintained with 70% nitrous oxide/30% oxygen and sevofluorane. Neuromuscular blockade will be obtained with rocuronium bromide 0.6 mg/kg.

After complete muscle paralysis (train of four = 0), the allocated SAD will be inserted by the study anesthesiologist according to the manufacturer's instructions.

The time to effective SGAD insertion will be define by the time between the devices was in the level of the lip patients until the CO2 waveform will be observed on the monitor display.

When more than one insertion attempt will be require, the patient will be receive bag-and-mask ventilation between attempts. A fail insertion attempt will be defined as complete withdrawal of the device from the mouth following an unsuccessful placement.

After two attempts the device will be deemed to have fail and the study protocol will be stop.The treating anesthetesiologist will then proceeded with the airway management of their choosing according to the needs of the patient and the surgery.

After achieving satisfactory ventilation via the allocated SAD, fibreoptic-guided tracheal intubation will be start.

A fiberscope (Karl Storz, Tuttlingen, Germany) with an outer diameter of 4.8 mm was used in all fiberoptic-guided procedures. All intubations will be perform with a disposable Endotracheal Tube with a low pressure, high volume cuff (VBM Medizintechnik GmbH, Sulz, Germany) with an internal diameter of 7.5 mm.

The flexible fiberscope will be loaded with the tracheal tube (TT), and advanced 2 cm beyond the TT for guidance. The participant will advance the fiberscope to the end of the SAD and the glottis will be view and assessed.

The scope will be insert into the trachea, the ETT will be railroad into the trachea, and the fibrescope will be then remove. Proper placement of the ETT will be confirm clinically and by the presence of the end tidal CO2 trace. The SAD will be then removed according to the manufacturer's instructions. After this maneuver the position of the ETT relative to the carina will be assessed bronchoscopicaly.

A maximum of two attempts will be s allowed with fibreoptic guided intubation. An alternative airway management plan could be instituted at the criterion by the anesthesiologist if a failed intubation is encountered after two attempts with the allocated device. The time of fiberscope intubation will be defined how the time when the fiberoscope is inserted in the ventilation channel of the SGAD until the presence of the CO2 waveform trace in the display of the monitor.

The primary outcome variable will be the total time to achieve successful fibreoptic intubation through the SADs (time to insertion of the SAD plus time to fibreoptic TI). Secondary variables included the following: SAD insertion time; TT insertion time; intubation success rate, and glottic view according to the Fiber-Optic Scoring System proposed by Brimacombe et al. In order to standardize the assessment of the SGD position (4 = only vocal cords seen; 3 = vocal cords plus posterior epiglottwill be seen; 2 = vocal cords plus anterior epiglottis seen; 1= vocal cords not seen), maneuvers performed to achieve TI (up-down mobilization or side to side mobilization) and Likert scale.

The anesthesiologist will be asked to rate the ease of use of the fiberscope-guided technique on a Likert scale for each technique, using the statement: ''The TT was easily inserted into the trachea'' (1 = strongly agree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree, 5 = strongly agree) (8).

Statistical analysis will be performed. The primary outcome will be time to fiberoptic-guided TI. Based on the pilot study, the investigator expected to obtain a large Cohen's d effect size corresponding to a time difference of at least 10 s, relative to the observed standard deviations (SDs) (9). In order to achieve a statistical significance for such mean time differences when using a repeated-measures procedure with an overall significance level of 0.05 (a = 0.05/3 for each pair with the Bonferroni adjustment) and a power of 0.8, a sample size of 24 would be necessary. The statistical power was calculated using G*Power free, version 3.0.10 (Franz Faul, University of Kiel, Kiel, Germany). A repeated-measures model was used to compare the mean time measurements (SAD insertion time, time to TI, and total time to secure the airway using fiberscope intubation technique among the two devices.

Categorical data were analyzed with nonparametric Friedman's two-way analysis of variance test. If the results were statistically significant at a 5% significance level, the tests were followed by post-hoc multiple compare between each pair of study devices. The paired t-test was used to analyze continuous data, and the Sign test was used to compare two dependent samples of categorical data sets.

According to Bonferroni multiple comparison adjustments, when comparing each pair of devices, p values <0.017 were considered statistical significant. SPSS, version 20 (SPSS Inc., IBM Corp.) was used for statistical analysis be. Continuous data will be presented as mean (SD). Categorical data will be presented as n (%)

ELIGIBILITY:
Inclusion criteria:

1. Patients with normal airway
2. weight 50-90kg
3. AGE 18-75
4. ASA I-II

Exclusion criteria:

1. predicted difficult airway
2. weight > 90 Kg
3. aspiration risk
4. pregnancy woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit patients if they are ≥18 years of age and of American Society of Anesthesiologists (ASA) physical status 1-2
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
time of success fiberoptic endotracheal intubation | 60 seconds
  seconds

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, M.D., Study Director — Bnai Zion Medical Center Haifa Israel